CLINICAL TRIAL: NCT07051499
Title: Effectiveness of TAP Block Versus Intravenous Analgesia in Postoperative Pain Management Following Gynecological Laparoscopic Surgery
Brief Title: Effectiveness of TAP Block Versus Intravenous Analgesia in Postoperative Pain Management Following Gynecologic Laparoscopic Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Michela Rauseo, MD, PhD, University of Foggia
Other Study IDs: TAP BLOCK GYNECOLOGIC SURGERY
Record Dates: First submitted 2025-06-13; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Pain
Keywords: Gynecologic surgery; Pain management; TAP Block; Regional Anesthesia; Intravenous Analgesia; ERAS
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- tap block group: - TAP Block Group: Bilateral ultrasound-guided TAP block with 0.25% levobupivacaine and 75 mcg clonidine per side, plus standard intraoperative intravenous analgesia (ketorolac, tramadol, ondansetron).
- intravenous analgesia: Standard intraoperative intravenous analgesia as above, followed by a postoperative elastomeric pump delivering tramadol 500 mg and ondansetron in 100 ml saline at 2 ml/h for 48 hours.
  Interventions: Drug: TAP Block Group

INTERVENTIONS:
Drug: TAP Block Group — Bilateral ultrasound-guided TAP block with 0.25% levobupivacaine and 75 mcg clonidine per side, plus standard intraoperative intravenous analgesia (ketorolac, tramadol, ondansetron).
  Groups: intravenous analgesia

SUMMARY:
Optimal postoperative pain control is crucial in laparoscopic gynecologic surgery, particularly within Enhanced Recovery After Surgery (ERAS) protocols. The transversus abdominis plane (TAP) block is a regional anesthesia technique that may reduce opioid consumption and enhance recovery. However, data comparing TAP block directly with standard intravenous analgesia in this surgical context are limited.

DETAILED DESCRIPTION:
This prospective, randomized controlled trial included patients undergoing laparoscopic gynecologic procedures (e.g., myomectomy, ovarian cystectomy, endometriosis surgery). Patients were randomized into two groups:

* TAP Block Group: Bilateral ultrasound-guided TAP block with 0.25% levobupivacaine and 75 mcg clonidine per side, plus standard intraoperative intravenous analgesia (ketorolac, tramadol, ondansetron).
* Intravenous Analgesia Group: Standard intraoperative intravenous analgesia as above, followed by a postoperative elastomeric pump delivering tramadol 500 mg and ondansetron in 100 ml saline at 2 ml/h for 48 hours.

Primary outcome: Postoperative pain intensity (NRS) at 1, 6, and 24 hours. Secondary outcomes included additional analgesic use, side effects, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years, scheduled for elective gynecological surgery

Exclusion Criteria:

* age <18, emergency surgery

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — all consecutive women undergoing gynecological surgery
Study Population: patients undergoing laparoscopic gynecologic procedures (e.g., myomectomy, ovarian cystectomy, endometriosis surgery).
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-01-21 (Estimated); Study Completion 2026-01-21 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity (Numeric Rating Scale) | 1, 6, 24 hours postoperatively.
  Postoperative pain will be assessed using the 11-point Numeric Rating Scale (NRS), where 0 indicates no pain and 10 indicates the worst imaginable pain. Higher scores indicate worse pain. Pain scores will be recorded at 1, 6, and 24 hours postoperatively.

SECONDARY OUTCOMES:
Total Analgesic Consuption. | 0-24 hours postoperatively.
  Total dose of tramadol (in Milligrams) administered in the first 24 hours after surgery will be recorded and compared between groups.
Incidence of Side Effects. | 0-24 hours postoperatively
  Occurrence of side effects such nausea, vomiting and sedation will be recorded and expressed as a percentage of patients (%) affected in each group.
Patient Satisfaction With Analgesia | 24 hours postoperatively
  Patient satisfaction with postoperative pain management will be assessed using a 5-point Likert scale (1= very dissatisfied; 5= very satisfied) at 24 hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico di Foggia, Foggia, Apulia, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Not sure